CLINICAL TRIAL: NCT04664270
Title: Developing and Implementing an Online Psychotherapy Program to Address Mental Health Challenges in Oncology and Palliative Care
Brief Title: Developing and Implementing E-psychotherapy Program for Mental Health Challenges in Oncology and Palliative Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Nazanin Alavi (Other)
Collaborators: Online PsychoTherapy Clinic (Other)
Responsible Party: Sponsor-Investigator, Dr. Nazanin Alavi, Principal Investigator, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSIY-699-20
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Mental Health Issue; Depression; Anxiety; Palliative Care; Oncology
Keywords: Mental Health; Virtual Care; Depression; Anxiety; Palliative Care; Psychotherapy
MeSH Terms: conditions — Depression; Anxiety Disorders; Neoplasms; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Randomly allocated to either treatment or control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-Psychotherapy (Experimental): Group will receive 8-week online program including CBT in combination with mindfulness and problem-based therapy in addition to treatment as usual. The content will reflect challenges cancer and palliative patients face through the course of treatment and developed into interactive and engaging therapy modules. All online sessions and interactions will occur through a secure online platform. Pre-designed therapy modules are assigned to the patients, accessible to them at any time throughout the week. Each module consists of approximately 30 slides, which take 45-50 minutes to complete. Each module highlights a different topic and includes general information, an overview of skills, and homework that is to be completed within that week. This homework can be directly submitted through the platform to the clinician who will then provide personalized feed-back to the patient. The average time spent per week by a clinician with a particular patient is about 15 minutes.
  Interventions: Behavioral: e-CBT
- Treatment as Usual (No Intervention): The control group will receive treatment as usual in the first 8 weeks; if still significantly symptomatic (less than 50% response to treatment from baseline), they will then be offered the 8-week e-psychotherapy program. They will be instructed to continue with any lifestyle activities (i.e., diet, exercise, medication, etc.)

INTERVENTIONS:
Behavioral: e-CBT — e-CBT + Mindfulness + Problem Solving
  Arms: e-Psychotherapy

SUMMARY:
The demand for mental health problems, particularly depression and anxiety, is three times greater in Oncology and Palliative Care Centres than in the general population. There are unique factors in this population that make them more susceptible to mental health challenges. The disease itself, the adjustment to a chronic/fatal diagnosis, and the treatment options can all perpetuate the development of mental illness. Despite the well-established association, there have been barriers to access suitable treatment for these patients.

Online Psychotherapy is an effective treatment option that may address many of these barriers. This modality has been proven effective in addressing depression and anxiety in other populations. To date, there has been no psychotherapy module developed specifically for oncology and palliative care patients to our knowledge. The aim is to establish the first academic e-psychotherapy treatment option to address mood and anxiety disorders in oncology and palliative care patients. The investigators will use the Online Psychotherapy Tool (OPTT), a secure cloud-based platform for online delivery of e-CBT, developed by the PI.

The proposed study aims to establish the feasibility and effectiveness of delivering online psychotherapy to oncology and palliative care patients who have a comorbid depressive or anxiety disorder. The patients will be enrolled in an 8-week program with a combination of cognitive behavioural therapy (CBT) and Mindfulness techniques delivered via a series of modules. They will receive individualized feedback from a trained therapist weekly. It is hypothesized that delivering this psychotherapeutic intervention in this manner will have great adherence. The aim is to prove that it will improve the quality of life and decrease symptoms of depression and anxiety in this underserved patient population.

DETAILED DESCRIPTION:
Sixty patients (n=60) diagnosed with depressive or anxiety disorder due to another medical condition in the context of cancer or palliative care, will be recruited to the study through referrals from health care professionals at Kingston Health Sciences Centre (KHSC) including cancer centre, Providence Care Hospital (PCH), family physicians, and other health care providers or self-referrals. After consenting to take part in the study, a complete assessment will be done by one of the psychiatrists on the team to confirm the diagnosis. Inclusion criteria include 18-55 years of age at the start of the study, diagnosed with depression or anxiety secondary to a general medical condition (in the context of cancer or palliative condition) according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) by one of the psychiatrists on the team, competence to consent and participate, ability to speak and read English, and consistent and reliable access to the internet. Exclusion criteria include acute hypomanic/manic episodes, acute psychosis, severe alcohol or substance use disorder, and active suicidal or homicidal ideation or if they have received CBT in the past year or are currently receiving CBT. Participants will then be randomly assigned to two groups: e-psychotherapy group (online CBT+ mindfulness + problem solving) or treatment as usual (TAU, i.e., medication, psychiatric consultation and referrals to in-person activities/groups) arms of the study (n=30 for each group). The TAU arm acts as the control group of the study.

Upon completion of the initial assessment, if eligible for the study, participants will randomly be assigned to one of the two arms of the study. Patients in the e-CBT group will receive an 8-week online program including CBT in combination with mindfulness and problem-based therapy in addition to treatment as usual. The content of this program will be customized to reflect challenges cancer and palliative patients face through the course of their treatment and developed into interactive and engaging therapy modules. All online sessions and interactions will occur through a secure online platform (i.e. OPTT). Through the platform, the pre-designed therapy modules are assigned to the patients, accessible to them at any time throughout the week. Each module consists of approximately 30 slides, which take an average of 45-50 minutes to complete. Each weekly module highlights a different topic and includes general information, an overview of skills, and homework that is to be completed within that week. This homework can be directly submitted through the platform to the clinician who will then provide personalized feed-back to the patient. The average time spent per week by a clinician with a particular patient is about 15 minutes. The control group will receive treatment as usual in the first 8 weeks; if still significantly symptomatic (less than 50% response to treatment from baseline), they will then be offered the 8-week e-psychotherapy program.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with depressive or anxiety disorder due to another medical condition in the context of cancer or palliative care
* competence to consent and participate
* speak and read English
* consistent and reliable access to the internet

Exclusion Criteria:

* acute hypomanic/manic episodes
* acute psychosis
* severe alcohol or substance use disorder
* active suicidal or homicidal ideation
* received CBT in the past year or are currently receiving CBT

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in symptoms (Functional Assessment of Cancer Therapy General - FACT-G) | Baseline, week 4, week 8
  Clinically validated symptom questionnaire. Scale of 0-4, 4 is worse.
Change in symptoms (Patient Health Questionnaire - PHQ-9 Item) | Baseline, week 4, week 8
  Clinically validated symptom questionnaire. Scale of 0-3, 3 is worse.
Change in symptoms (Generalized Anxiety Disorder - GAD7 Item) | Baseline, week 4, week 8
  Clinically validated symptom questionnaire. Scale of 0-3, 3 is worse.
Change in symptoms (Quality of Life and Satisfaction Questionnaire - Q-LES-Q) | Baseline, week 4, week 8
  Clinically validated symptom questionnaire. Scale of 0-5, 5 is better.

SECONDARY OUTCOMES:
Changes in frequency on online platform | Week 8
  Logins per day
Changes in duration on online platform | Week 8
  Amount of time spent on each session

CONTACTS AND LOCATIONS:
Overall Officials: Nazanin Alavi, Principal Investigator — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

REFERENCES:
- [Derived] Alavi N, Stephenson C, Miller S, Khalafi P, Sinan I, Kain D, McDougall M, Davies J, Stark D, Tompkins E, Jagayat J, Omrani M, Shirazi A, Groll D, Soares C. Developing and Implementing a Web-Based Psychotherapy Program to Address Mental Health Challenges Among Patients Receiving Oncologic and Palliative Care: Protocol for an Open-Label Randomized Controlled Trial. JMIR Res Protoc. 2021 Jul 14;10(7):e30735. doi: 10.2196/30735. PMID 34259164